CLINICAL TRIAL: NCT03171623
Title: A Randomised,Double-blind,Placebo-controlled Study to Assessment of Single-Dose Safety,Tolerability, Pharmacokinetics and Pharmacodynamic of Globalagliatin Hydrochloride (SY-004) in Chinese Healthy Subjects
Brief Title: The Assessment of Single-Dose Safety,Tolerability, Pharmacokinetics and Pharmacodynamic of Globalagliatin Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yabao Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YB002003
Record Dates: First submitted 2017-05-05; First posted 2017-05-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Hyperglycaemia (Diabetic); Healthy Volunteers
Keywords: T2DM; Diabetes; GKA
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SY-004 2mg (Experimental): SY-004 (globalagliatin hydrochloride) 2mg by mouth, single dose
  Interventions: Drug: globalagliatin hydrochloride
- SY-004 20mg&placebo (Placebo Comparator): SY-004 (globalagliatin hydrochloride) 20mg or placebo by mouth, single dose
  Interventions: Drug: globalagliatin hydrochloride; Drug: placebo
- SY-004 40mg&placebo (Placebo Comparator): SY-004 (globalagliatin hydrochloride) 40mg or placebo by mouth, single dose
  Interventions: Drug: globalagliatin hydrochloride; Drug: placebo
- SY-004 80mg&placebo (Placebo Comparator): SY-004 (globalagliatin hydrochloride) 80mg or placebo by mouth, single dose
  Interventions: Drug: globalagliatin hydrochloride; Drug: placebo
- SY-004 120mg&placebo (Placebo Comparator): SY-004(globalagliatin hydrochloride) 120mg or placebo by mouth, single dose
  Interventions: Drug: globalagliatin hydrochloride; Drug: placebo

INTERVENTIONS:
Drug: globalagliatin hydrochloride — orally administration, single dose
  Other Names: SY-004 capsule
Drug: placebo — orally administration, single dose
  Arms: SY-004 120mg&placebo; SY-004 20mg&placebo; SY-004 40mg&placebo; SY-004 80mg&placebo

SUMMARY:
This is a phase 1 randomized,double-blind,placebo-controlled study with single oral dose of globalagliatin hydrochloride (SY-004) administered to chinese healthy subjects to evaluated the safety, tolerability, pharmacokinetics and pharmacodynamics of globalagliatin hydrochloride (SY-004).

DETAILED DESCRIPTION:
Glucokinase is a characteristic hexokinase isoenzyme in hepatocytes that catalyzes the first step in glucose metabolism. In addition to its role in glucose metabolism, glucokinase is expressed in pancreatic islet beta cells where it acts as a "glucose sensor" for insulin release. Activation of glucokinase increases the glucose sensitivity of insulin secretion, effectively lowering the glucose threshold for insulin secretion. Because of its potential to enhance insulin secretion and affect hepatic glucose metabolism, is being investigated for use as a treatment for hyperglycaemia,glubalagliatin( the active ingredient in SY-004 capsule) is being investigated for use as a treatment for T2DM patients. This is a phase 1 randomized,double-blind,placebo-controlled study with single oral dose of SY-004 administered to chinese healthy subjects to evaluated the safety, tolerability, pharmacokinetics and pharmacodynamics of SY-004.

ELIGIBILITY:
Inclusion Criteria:

* males and females between the ages of 18 and 65 years, inclusive, healthy subjects
* A screening body mass index (BMI) of 18 to 26 kg/m2 inclusive, body weight above 50kg
* FPG≥3.9mmol/L and <6.1 mmol/L
* Have medical history, physical examination, laboratory tests and other relative test results within the normal range or with abnormalities deemed clinically insignificant by the investigator.
* Have given written informed consent.
* The subjects took effective contraceptive measures, and had no birth plan within 3 months.Female subjects should be non lactating, negative pregnancy test, or no fertility potential (Women who were 12 months of menopause or without uterus were found to have no potential for pregnancy )

Exclusion Criteria:

* There is a serious history of systemic disease, or a family history (including cardiovascular system, digestive system, urinary system, etc.)
* Have taken a special diet or exercise before 48 hours of drug administration or other factors are capable of significantly altering the absorption, or metabolism or elimination of drugs.
* A significant abnormality in ALT,AST or other lab test results
* Frontal chest X light result is clinical significantly abnormal.
* Have known intolerance of or allergies to glucokinase activators, or related compounds.
* Have known allergies to other compounds or biologic products.
* Have a major surgery in the last 4 weeks before dosing.
* To inoculate any live vaccine within 4 weeks before drug administration.
* Have a history of drug abuse
* Use any prescription drugs within 4 weeks prior to administration or use OTC or traditional Chinese medicine within 1 weeks before enrollment.
* Regular drinkers within 6 months before or during the trial (Subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) [1 unit = 360 mL of beer; or 150 mL of wine; or 45 mL of distilled spirits])
* The amount of daily cigarette smoking was more than 5/day in last 3 months, or subjects unwilling to stop cigarette consumption during the trial.
* Are enrolled in 4 or more clinical trials within last year, or participated any clinical trail within 3 months before enrollment ; plan to donate blood or blood donation of 450 mL or more in the last 3 months; or have blood transfusion 4 weeks before the trial.
* An clinical significant abnormality in the 12-lead ECG at screening or baseline: QT interval> 450 ms
* Subjects deemed unsuitable by the Investigator for low compliance or any other reason.
* investigator and their immediate families.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single dose of SY-004 | 14 day post-dose
  number of patients with adverse events and changes from baseline in vital signs, ECG and clinical labs (blood chemistry, hematology and urinalysis)

SECONDARY OUTCOMES:
AUC of SY-004 following oral administration of single ascending dose | up to 168 hours post-dose
  to measure the study drug concentration in blood and urine samples to be collected after drug administration.
Cmax of SY-004 following oral administration of single ascending dose. | up to 168 hours post-dose
  to measure the study drug concentration in blood and urine samples to be collected after drug administration.
T1/2 of SY-004 following oral administration of single ascending dose | up to 168 hours post-dose
  to measure the study drug concentration in blood and urine samples to be collected after drug administration.
CL/F of SY-004 following oral administration of single ascending dose | up to 168 hours post-dose
  to measure the study drug concentration in blood and urine samples to be collected after drug administration.
glucose levels following single dose of SY-004 | up to 48 hours post-dose
  FPG AUC
insulin secretion following single dose of SY-004 | up to 11 hours post-dose
  insulin changes
C-peptide secretion following single dose of SY-004 | up to 11 hour post-dose
  C-peptide change

CONTACTS AND LOCATIONS:
Overall Officials: Lei Yang, Study Director — Yabao pharmaceutical Group Co.
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao Y, Xie L, Zhang H, Zhou S, Liu Y, Chen J, Wang L, Wang L, Zhuo L, Wang Y, Ou N, Shao F. Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of SY-004, a Glucokinase Activator, in Healthy Chinese Adults: A Randomized, Phase Ia, Single-Ascending Dose Study. Clin Ther. 2022 Feb;44(2):269-281. doi: 10.1016/j.clinthera.2021.12.009. Epub 2022 Jan 29. PMID 35093240